CLINICAL TRIAL: NCT06918717
Title: Assessment of Prehospital Tracheal Intubation Technique Using Initial Direct Laryngoscopy During Videolaryngoscopy: Randomized Controlled Simulated Trial
Brief Title: Prehospital Tracheal Intubation Technique Using Initial Direct Laryngoscopy During Videolaryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Cédric Cibotto, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Req-2023-00073
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Tracheal Intubation
Keywords: Advanced airway management; direct laryngoscopy; tracheal intubation; prehospital; videolaryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free use of videolaryngoscopy (Active Comparator)
  Interventions: Procedure: Free use of videolaryngoscopy
- Direct Laryngoscopy-to-VideoLaryngoscopy sequence (Experimental)
  Interventions: Procedure: Direct Laryngoscopy-to-VideoLaryngoscopy sequence

INTERVENTIONS:
Procedure: Direct Laryngoscopy-to-VideoLaryngoscopy sequence — Participants will proceed with a double intubation technique sequence, first performing an initial direct laryngoscopy without looking at the video screen until they reached the epiglottis, then performing an indirect lryngoscopy for intubation.
  Arms: Direct Laryngoscopy-to-VideoLaryngoscopy sequence
Procedure: Free use of videolaryngoscopy — Participants are free to use of the videolaryngoscope as they intended
  Arms: Free use of videolaryngoscopy

SUMMARY:
Tracheal intubation using videolaryngoscopy may be required in the prehospital setting, where airway management presents unique technical and logistical challenges. Intubation may be hard because novice providers performing videolaryngoscopy may only look at the screen and only obtain a two-dimensional representation of the patient's airways. By directly visualizing the airways, these providers may obtain a better 3D apprehension and an improved mental visualization of the patient's anatomy. We aim to compare the impact of a freely realized videolaryngoscopy sequence with a sequence consisting in direct visualization of the airway followed by videolaryngoscopy ("Direct Laryngoscopy-to-VideoLaryngoscopy sequence" or "DL-VL sequence") on time to intubation among novice providers.

ELIGIBILITY:
Inclusion Criteria:

* All resident physicians with 1 to 6 years of post-graduate experience working in the Emergency Department (ED) at Geneva University Hospitals (Hôpitaux Universitaires de Genève (HUG)) and penultimate year of medical school students (5th year) studying at University of Geneva Faculty of Medicine (UGFM).
* Performed less than 10 ETIs prior to participating in the study.

Exclusion Criteria:

* More than 6 years of post-graduate experience
* Performed more than 10 ETIs prior to participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Time to Intubation | Periprocedural
  Time in seconds from blade insertion at the dental arch to adequate tracheal tube placement through the vocal cords, confirmed by the C-MAC video recording. A maximum of 60 seconds was allowed per ETI attempt. The maximum number of ETI attempts was limited to 3.

SECONDARY OUTCOMES:
Time to Intubation for the first intubation attempt alone | Periprocedural
  Time in seconds from blade insertion at the dental arch to adequate tracheal tube placement through the vocal cords, confirmed by the C-MAC video recording. A maximum of 60 seconds was allowed per ETI attempt.
First Pass Success rate | Periprocedural
  Intubation first pass success rate, in percentage.
Number of intubations attempts | Periprocedural
  An ETI attempt was defined as the insertion of the laryngoscope blade at the dental arch, regardless of whether tracheal tube placement was attempted. A maximum of 60 seconds was allowed per ETI attempt. The maximum number of ETI attempts was limited to 3. More than 3 attempts, it was considered as failed.
Time to Ventilation | Periprocedural
  Time in seconds from blade insertion at the dental arch to successful ventilation confirmed by chest elevation. A maximum of 60 seconds was allowed per ETI attempt.
Subjective assessments | Periprocedural
  Subjective assessments, including perceived difficulty (Question 1 - I found intubation easy. Question 2 - I felt comfortable intubating this way. Question 3 - I think the use of the VL was adequate to intubate OR I think the sequenced use of the VL helped me intubate. Question 4 - In a future similar clinical situation, I will make the same use of the VL to intubate OR I think doing a direct laryngoscopy before looking at the screen allows for faster intubation than doing an indirect laryngoscopy only. Question 5 - In a future similar clinical situation, I will make a different use of the VL to intubate OR In a future similar clinical situation, I will make the same use (DL-VL) of the VL to intubate. Question 6 - In a future similar clinical situation, I will make a different use (VL only) of the VL to intubate.), were appraised using a 5-point Likert scale ranging from "Totally Agree" to "Totally Disagree".

CONTACTS AND LOCATIONS:
Overall Officials: PD Dr Laurent Suppan, Study Director — University Hospital, Geneva
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Cibotto C, Pasquier M, Beysard N, Rouyer F, Grosgurin O, Bourgeois L, Erriquez E, Braun E, Gartner BA, Desmettre T, Suppan L. Assessment of prehospital tracheal intubation technique using initial direct laryngoscopy during videolaryngoscopy: randomized controlled simulated trial. BMC Emerg Med. 2025 Jul 1;25(1):112. doi: 10.1186/s12873-025-01266-0. PMID 40596822